CLINICAL TRIAL: NCT00001548
Title: Genetics of Obsessive-Compulsive Disorder: A Collaborative Study
Brief Title: Genetics of Obsessive-Compulsive Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960124; 96-M-0124
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-09-29

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Genetic; Psychiatric Disorder; Affected Sib Pairs; Obsessions; Compulsions; Family Study; OCD Spectrum Disorders; Trichotillomania; Tourette's Syndrome
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Mental Disorders; Obsessive Behavior; Compulsive Behavior; Trichotillomania; Tourette Syndrome

SUMMARY:
The purpose of this study is to identify genes that affect susceptibility to obsessive-compulsive disorder (OCD). By identifying genes that increase or decrease the risk of OCD, researchers can better understand how the condition develops and ultimately improve treatment for people with OCD.

OCD is a severe, familial condition that affects approximately 2% of the population. The way OCD is inherited is not clearly understood, but researchers believe it is complex and involves multiple genes. This study will detect and localize genes that increase or decrease susceptibility to OCD. The data collected from this study will be combined with data from other research studies to determine gene linkage and association.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a severe, heritable condition with a lifetime prevalence of about two percent of the population. The mode of inheritance is poorly understood but is likely complex, involving multiple loci of small to major effect. Since 1995, the NIMH-IRP has been active in a multi-center family study of OCD, led by Dr. Gerald Nestadt of Johns Hopkins University, which was approved via a competitive NIMH extramural application (MH 502140). An expanded consortium of sites (including new sites at Brown and Harvard Universities) anticipates adding 300 new affected sib-pair families over the next three years. This sample will be used for linkage and association analyses. Data will be shared within this consortium of investigators studying OCD, and will eventually be combined with data obtained from a second consortium.

ELIGIBILITY:
* INCLUSION CRITERIA:

Must have a diagnosis of obsessive-compulsive disorder, or be a family member (usually a parent or sibling) of someone with obsessive-compulsive disorder.

Certain disorders are considered part of OCD "spectrum" disorders and often include family members with OCD. These include Tourette's Syndrome, other individuals with tics, and Trichotillomania (severe hair pulling), and other forms of repetitive behaviors.

Persons with primary behavioral difficulties who do not fit with the current definitions of "OCD and OCD spectrum disorders" may not be eligible. These include compulsive shopping, gambling, or compulsive sexual behaviors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 1996-08-22; Study Completion 2015-09-29

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McMahon, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wendland JR, Moya PR, Timpano KR, Anavitarte AP, Kruse MR, Wheaton MG, Ren-Patterson RF, Murphy DL. A haplotype containing quantitative trait loci for SLC1A1 gene expression and its association with obsessive-compulsive disorder. Arch Gen Psychiatry. 2009 Apr;66(4):408-16. doi: 10.1001/archgenpsychiatry.2009.6. PMID 19349310
- [Background] Zuchner S, Wendland JR, Ashley-Koch AE, Collins AL, Tran-Viet KN, Quinn K, Timpano KC, Cuccaro ML, Pericak-Vance MA, Steffens DC, Krishnan KR, Feng G, Murphy DL. Multiple rare SAPAP3 missense variants in trichotillomania and OCD. Mol Psychiatry. 2009 Jan;14(1):6-9. doi: 10.1038/mp.2008.83. No abstract available. PMID 19096451
- [Background] Wendland JR, Moya PR, Kruse MR, Ren-Patterson RF, Jensen CL, Timpano KR, Murphy DL. A novel, putative gain-of-function haplotype at SLC6A4 associates with obsessive-compulsive disorder. Hum Mol Genet. 2008 Mar 1;17(5):717-23. doi: 10.1093/hmg/ddm343. Epub 2007 Nov 30. PMID 18055562